CLINICAL TRIAL: NCT01998243
Title: Usefulness Of Intra-Gastric Balloon Before Bariatric Surgery In Morbid Obesity To Decrease Bariatric Surgery Morbidity
Brief Title: Usefulness and Safeness Of Intra-Gastric Balloon Before Bariatric Surgery In Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Severo Ochoa (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, luis ramon rábago torre, Dr. Phd Luis Ramon Rábago Torre, Hospital Severo Ochoa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fis PI070682; FIS PI070682 (Other Grant/Funding Number: SPANISH NATIONAL HEALTH SYSTEM, LAIN ENTRALGO AGENCY)
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; bioenterics intragastric balloon; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Drug Delivery Systems; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGB group A (Experimental): the intervention in the group A : was to place a preoperative intragastric balloon (IGB-BIB®) in the stomach for 6 months before surgery plus an hypocaloric diet 1200 Kilocalories (Kcal)
  Interventions: Device: Intragastric Balloon (IGB), group A; Other: diet, control group B
- control group B (Placebo Comparator): the intervention in this control group B was the specified diet (a hypocaloric diet of 1200 Kilocalories (Kcal)
  Interventions: Other: diet, control group B

INTERVENTIONS:
Device: Intragastric Balloon (IGB), group A — the intervention was to place An intragastric balloon (BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM) endoscopically under conscious sedation and was kept in the stomach during minimum 6 months. Patients were also treated with proton bomb inhibitors (PPI), and prokinetics to control gastroesophageal reflux . The balloon was endoscopically removed with the patient under general anesthesia to avoid bronco-aspiration related problems
  Other Names: BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM
  Arms: IGB group A
Other: diet, control group B — the intervention in this cotrol group B was only 1200 Kilocalories (Kcal) diet
  Other Names: 1200 Kilocalories (Kcal) diet

SUMMARY:
Introduction: bariatric surgery shows an important morbidity and there are some reports that have used preoperative intragastric-balloons (IGB-BIB®) to decrease surgical morbidity.

Patients Methods: Since 2009 we are performing a randomized and prospective study to assess the usefulness of (IGB-BIB®) before bariatric surgery [sleeve resection (SR) or gastric bypass (GB)] "group A". The intervention in this group was was to place an intragastric Balloon for 6 months vs a control group "B" with the same type of surgical procedures but without preoperative IGB-BIB.The intervention on this group was only to treat the obesity only with diet for 6 months . All patients coming for both groups were followed at 4-week intervals by a nurse practitioner and dietitian for 6 months, Nurse practitioner made the dietetics adjustments (750-1500 Kcal) , provide advice and assess the evolution of weight loss The hypothesis was that preoperative IGB-BIB helps the patients to lose weight ( more than 10%) ,and the weight loss will contribute to decrease surgical morbidity by at least 30%, and also will decrease hospital stay Objective: to check if morbidity, mortality and hospital stay decreased in the IGB-BIB ® group, and secondly if the weight before surgery was associated with surgical morbidity. secondary objective : Assess the rate of IGB-BIB failure.Intragastric balloon failure was considered when the weight loss is less than 10% from the initial weight. We defined severe complication whenever the patient had to be admitted in the hospital after discharge, new surgeries or transfusions were required or the hospital stay was longer than 7-10 days.

DETAILED DESCRIPTION:
Treatment with an intragastric balloon (IGB) for morbid obesity is a temporary treatment reached as a second step, when the initial nutritional multidisciplinary approach has failed; however, its value is not clear compared with other conventional medical treatments ], though some authors have stated that IGB achieves higher weight loss than conventional diet treatments (12.2% of the initial weight) ]; and others have positioned IGB as the first valid step in order to achieve weight loss in patients who are adequate for a future gastric bypass surgery. Genco et al (2009) have compared the treatment with IGB only vs. laparoscopic sleeve gastrectomy (LSG), and have found no differences in the amount of weight loss at 6 months, but a reduction in adverse events caused by IGB treatment.

One of the potential future indications for the intragastric balloon could be its use as a bridge-treatment until bariatric surgery, not only in order to achieve weight loss before surgery, but also to select the group of patients who might benefit more from derivative surgery, as suggested by some authors or its use in special populations such as super-obese patients . The objective would be to reduce weight before the surgical procedure, in order to improve comorbidities, facilitate the surgical technique, and potentially reduce any surgical complications.

It is increasingly frequent in many surgical units to try and achieve weigh loss before bariatric surgery, using intragastric balloons (IGB). However, this therapeutic approach currently presents dubious utility. Our study intends to contribute with our experience in the evaluation of IGB before surgery for achieving weight loss, and its impact on post-surgical morbidity.

Bariatric surgery shows an important morbidity and there are not to many randomized prospective studies using intragastric- balloons (IGB-BIB®) to evaluate if getting weight lost really matter on decreasing surgical complications before Bariatric surgery OBJECTIVE: To study the usefulness of preoperative IGB-BIB® "grA" [sleeve resection (SR) or gastric bypass (GB)] to help decrease postsurgical complications. Secondly we try to check the rate of IGB-BIB® failures (a total weight loss less than 10% of the initial weight), and the impact on decreasing hospital stay and rate of surgical reoperations. METHODS: The study was a clinical prospective and randomized essay coming from 2009. Cases (grA) had an IGB during 6 months before surgery vs Controls (grB)

ELIGIBILITY:
Inclusion Criteria:

1. - Morbid obesity (BMI ≥ 40 kg/m2 ) with a failed Conventional Medical treatment
2. - Morbid obesity (BMI ≥ 35 kg/m2) with important comorbidity with a failed Conventional Medical treatment
3. - they should be operated by a laparoscopic gastric sleeve or by laparoscopic gastric by-pass

Exclusion Criteria:

1. - Slight adherence to previous medical treatments .
2. - Hiatal hernia more than 3 cms
3. - Patients with active gastric or duodenal ulcer disease
4. - Severe esophagitis
5. - Psychiatric diseases (depression, bulimia etc)
6. - Associated Severe Systemic Disease not amenable to improve with weight loss
7. - Patients with Inflammatory bowel diseases
8. - Patients on anticoagulant treatment or steroids .
9. - Addiction to Drugs or alcohol
10. - Past history of gastric surgery ,antireflux surgery or any other type of bariatric surgery
11. - Patient refusing to be followed 6 months before and after surgery
12. - Pregnancy or foreseeable pregnancy during the study
13. - Patients with gastric or esophageal varices
14. - proton pump inhibitor (PPI) allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis R Rábago, MD,PhD, Principal Investigator
Locations (1):
- Gastroenterology Department ,Severo Ochoa Hospital, Leganés, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodson RM, Zacharoulis D, Goutzamani E, Slee P, Wood S, Wedgwood KR. Management of obesity with the new intragastric balloon. Obes Surg. 2001 Jun;11(3):327-9. doi: 10.1381/096089201321336692. PMID 11433910
- [Background] Loffredo A, Cappuccio M, De Luca M, de Werra C, Galloro G, Naddeo M, Forestieri P. Three years experience with the new intragastric balloon, and a preoperative test for success with restrictive surgery. Obes Surg. 2001 Jun;11(3):330-3. doi: 10.1381/096089201321336700. PMID 11433911
- [Background] Doldi SB, Micheletto G, Perrini MN, Librenti MC, Rella S. Treatment of morbid obesity with intragastric balloon in association with diet. Obes Surg. 2002 Aug;12(4):583-7. doi: 10.1381/096089202762252398. PMID 12194556
- [Background] Busetto L, Segato G, De Luca M, Bortolozzi E, MacCari T, Magon A, Inelmen EM, Favretti F, Enzi G. Preoperative weight loss by intragastric balloon in super-obese patients treated with laparoscopic gastric banding: a case-control study. Obes Surg. 2004 May;14(5):671-6. doi: 10.1381/096089204323093471. PMID 15186637
- [Background] Sallet JA, Marchesini JB, Paiva DS, Komoto K, Pizani CE, Ribeiro ML, Miguel P, Ferraz AM, Sallet PC. Brazilian multicenter study of the intragastric balloon. Obes Surg. 2004 Aug;14(7):991-8. doi: 10.1381/0960892041719671. PMID 15329191
- [Background] Alfalah H, Philippe B, Ghazal F, Jany T, Arnalsteen L, Romon M, Pattou F. Intragastric balloon for preoperative weight reduction in candidates for laparoscopic gastric bypass with massive obesity. Obes Surg. 2006 Feb;16(2):147-50. doi: 10.1381/096089206775565104. PMID 16469215
- [Derived] Vicente Martin C, Rabago Torre LR, Castillo Herrera LA, Arias Rivero M, Perez Ferrer M, Collado Pacheco D, Martin Rios MD, Barba Martin R, Ramiro Martin J, Vazquez-Echarri J, Herrera Merino N. Preoperative intragastric balloon in morbid obesity is unable to decrease early postoperative morbidity of bariatric surgery (sleeve gastrectomy and gastric bypass): a clinical assay. Surg Endosc. 2020 Jun;34(6):2519-2531. doi: 10.1007/s00464-019-07061-w. Epub 2019 Aug 9. PMID 31399943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 patients were eligibles for the study and were evaluated at the endocrinologist office
Pre-assignment Details: 40 patients rejected to be included in the study and 30 were excluded before randomization for not to fulfill all the established requirement to be included
Groups:
- Group B: 42 patients control group : patients were followed during at least 6 months before surgery by the same group of nutritionist that followed the group A and with the same type of diet and diet recommendations
- IGB-BIB® Group A: 39 patients included have a preoperative intragastric balloon during a period of 6 months before operation
  preoperative intragastric balloon ( IGB-BIB®): An intragastric balloon (BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM)is placed endoscopically under conscious sedation was kept in the stomach during minimum 6 months. Patients were also treated with proton bomb inhibitors, and prokinetics to control gastroesophageal reflux . The balloon was endoscopically removed with the patient under general anesthesia to avoid bronco-aspiration related problems
Period: Overall Study
Arm/Group | Group B | IGB-BIB® Group A
Started | 42 | 39
Completed | 34 | 32
Not Completed | 8 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group B: this is the control group, It includes patients followed during at least 6 months before bariatric surgery by the same group of nutritionist that followed the group A and with the same type of diet and diet recommendations
- Intragastrc Balloon (IGB) Group A: this is the intervention group, it includes patients who had a preoperative intragastric balloon during a period of 6 months before operation
  preoperative intragastric balloon ( IGB-BIB®): An intragastric balloon (BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM)is placed endoscopically under conscious sedation was kept in the stomach during minimum 6 months. Patients were also treated with proton bomb inhibitors, and prokinetics to control gastroesophageal reflux . The balloon was endoscopically removed with the patient under general anesthesia to avoid bronco-aspiration related problems
- Total: Total of all reporting groups
Arm/Group | Group B | Intragastrc Balloon (IGB) Group A | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years OF AGE] | 42.6 (9.2) | 43 (10.2) | 42.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 32 | 66
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 34 | 32 | 66
Americam Society of Anestesiologist Physical Status Classification System (ASA) ; ASA score III; [Number; unit: participants] — Physical Status Classification System (ASA) ASA classification scores patients ranging from I - V ; ASA I A normal healthy patient Healthy, ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation E , ASA VI A declared brain-dead patient whose organs are being removed for donor purposes .WE MEASURE THE NUMBER of participants IN EACH GROUP classified as ASA III
  participants | 11 | 12 | 23
Starting weight (kg) [Mean (Standard Deviation); unit: Kg] — the starting weight is expressed in Kg
  Kg | 125 (18.5) | 129.2 (19.4) | 127.1 (18.9)
Starting body mass index (starting BMI) [Mean (Standard Deviation); unit: "kg/m^2"] — Starting body mass index (starting BMI) is expressed in kg/m^2
  "kg/m^2" | 46 (4.9) | 46.4 (6.9) | 46.2 (5.7)
Starting body mass index (starting BMI) > 50 ("kg/m^2") [Count of Participants; unit: Participants] — number of patientes with a Starting body mass index (starting BMI) > 50 "kg/m^2"
  Participants | 8 | 7 | 15
Total weight loss (TWL) [Median (Inter-Quartile Range); unit: Kg] — Total weight loss (TWL) is expressed in Kg
  Kg | 3 [1 to 6.5] | 16 [8.2 to 22.7] | 7 [3 to 17.7]
Weight before surgery (Kg) [Mean (Standard Deviation); unit: Kg] — Weight before surgery is expressed in KG
  Kg | 121.3 (20.5) | 112.8 (16.4) | 117.2 (19.0)
BMI before surgery("kg/m^2") [Mean (Standard Deviation); unit: "kg/m^2"] | 44.3 (5.5) | 40 (6.2) | 42.2 (5.9)
Excess weight loss (EWL) before surgery [Median (Inter-Quartile Range); unit: percentage of EWL] — Excess weight loss (EWL) before surgery is expressed as a percentage % Population: missing data
  percentage of EWL
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 4.54 [1.4 to 10.07] | 27.14 [12.2 to 35.2] | 11.1 [3.4 to 28.9]
Excess Body Mass Index Loss (EBMIL) before surgery (excess BMI loss) [Median (Inter-Quartile Range); unit: percentage of EBMI loss] | 1 [0 to 2] | 6.04 [3.9 to 7.9] | 3 [1 to 6.5]
Surgery (sleeve resection (LSG)or gastric bypass (LGBP) [Count of Participants; unit: Participants]
  LSG | 11 | 9 | 20
  LGBP | 23 | 23 | 46
total body weight loss (TBWL) > 10% [Count of Participants; unit: Participants] — Population: missing data
  Participants
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 4 | 18 | 22
Percentage of Failure of Intragastric Balloon [Count of Participants; unit: Participants] — It was considered that intragastric balloon failed when a total weight loss = or > than 10% of the starting weight has NOT been achieved.
  The total number of patients with IGB balloon was 41 in this essay, but 9 were excluded post randomization of the final analysis because they were not finally operated.
  The percentage of IGB balloon failure was calculated for all the patients had intragastric balloon Population: this variable is not applicable to group B
  Participants
    number analyzed (Participants) | 0 | 32 | 32
    (all) |  | 11 | 11
Operation time (hours) [Mean (Standard Deviation); unit: hours] — Operation time is expressed in hours Population: missing data
  hours
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 2.8 (0.73) | 2.8 (0.79) | 2.8 (0.76)
ICU (hours) intensive care unit [Median (Inter-Quartile Range); unit: hours)] — time spent in the intensive care unit is expressed in ICU (hours) Population: missing data
  hours)
    number analyzed (Participants) | 33 | 32 | 65
    (all) | 21.5 [7.2 to 23] | 11 [8 to 24] | 20 [8 to 23]

OUTCOME MEASURES:

1. Primary Outcome: Postsurgical Morbidity on Both Arms of the Study
Description: postsurgical morbidity includes all kind of post operative morbidity( mild ,moderate and severe) moderate and severe post surgical morbidity is the most important one
Time Frame: within the 90 days after surgery
Measure: Count of Participants; unit: Participants
Groups:
- IGB Group A: this is the intervention group, it includes patients who had a preoperative intragastric balloon during a period of 6 months before operation
  preoperative intragastric balloon ( IGB-BIB®): An intragastric balloon (BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM)is placed endoscopically under conscious sedation was kept in the stomach during minimum 6 months. Patients were also treated with proton bomb inhibitors, and prokinetics to control gastroesophageal reflux . The balloon was endoscopically removed with the patient under general anesthesia to avoid bronco-aspiration related problems
Arm/Group | Group B | IGB Group A
Number analyzed (Participants) | 34 | 32
Participants
  postsurgical morbidity | 10 | 8
  moderate-severe postsurgical morbidity | 8 | 4
Statistical Analysis 1: Comparison: Group B vs IGB Group A; Test type: Superiority; p = 0.689, Chi-squared; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.53 to 2.60] — risk ratio (RR)

2. Primary Outcome: Total Postsurgical Morbidity
Description: total postsurgical morbidity included the morbidity specifically due to the Intragastric balloon plus all the postoperative morbidity related to the surgical procedure severe intragastric balloon morbidity refers only to medical complications which meet the criteria of severe of "The accordion severity grading system ".
Time Frame: during the 6 months having the intragastric balloon and 90 days after surgery
Population: Group B did not receive an intra-gastric balloon, and was thus not evaluated for balloon related complications.
Measure: Count of Participants; unit: Participants
Groups:
- Group B: 34 patients control group : patients were followed during at least 6 months before surgery by the same group of nutritionist that followed the group A and with the same type of diet and diet recommendations
- IGB Group A: 32 patients included have a preoperative intragastric balloon during a period of 6 months before operation
  preoperative intragastric balloon ( IGB-BIB®): An intragastric balloon (BIOENTERICS INTRAGASTRIC BALLOON (BIB) SYSTEM)is placed endoscopically under conscious sedation was kept in the stomach during minimum 6 months. Patients were also treated with proton bomb inhibitors, and prokinetics to control gastroesophageal reflux . The balloon was endoscopically removed with the patient under general anesthesia to avoid bronco-aspiration related problems
Arm/Group | Group B | IGB Group A
Number analyzed (Participants) | 34 | 32
Participants
  intragastric balloon morbidity (complications): number analyzed (Participants) | 0 | 32
  intragastric balloon morbidity (complications) |  | 8
  severe intragastric balloon morbidity: number analyzed (Participants) | 0 | 32
  severe intragastric balloon morbidity |  | 2
  total postsurgical morbidity | 10 | 15
Statistical Analysis 1: Comparison: Group B vs IGB Group A; Test type: Superiority; p = 0.144, Chi-squared; Risk Ratio (RR) = 1.59, 95% CI 2-sided [0.84 to 3.01] — all in all balloon and postsurgical morbidity in group A vs. group B

3. Secondary Outcome: Hospital Stay,
Description: all in all hospital stay
Time Frame: the period of the study started when patients were randomizated and finished 90 days after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group B | IGB Group A
Number analyzed (Participants) | 34 | 32
days | 10.3 (15.3) | 7 (4.3)
Statistical Analysis 1: Comparison: Group B vs IGB Group A; Test type: Superiority; p = 0.937, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Rate of Surgical Conversion to Open Surgery
Description: number of patients with surgical conversion from laparoscopic to open surgery
Time Frame: during the initial laparoscopic surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group B | IGB Group A
Number analyzed (Participants) | 34 | 32
Participants | 1 | 1
Statistical Analysis 1: Comparison: Group B vs IGB Group A; Test type: Superiority; p = 1, Fisher Exact

5. Secondary Outcome: Percentage of Re-operations
Description: Percentage of Re-operations during all the period of the study ending within 90 days after surgery
Time Frame: during all the period of the study ending within 90 days after surgery
Measure: Number; unit: percentage of participants
Arm/Group | Group B | IGB Group A
Number analyzed (Participants) | 34 | 32
percentage of participants | 11.8 | 6.3
Statistical Analysis 1: Comparison: Group B vs IGB Group A; Test type: Superiority; p = 0.673, Fisher Exact

ADVERSE EVENTS:
Time Frame: from randomization six months before surgery to 90 days after surgey
Arm/Group | Group B | IGB Group A
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/34 | 1/32
Other Adverse Events (participants affected / at risk) | 8/34 | 7/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group B (N=34) | IGB Group A (N=32)
acute renal failure (Renal and urinary disorders) | 2 (8) | 1 (1) — peritonitis, sepsis, suture dehiscence, respiratory failure, eventration intraperitoneal postoperative bleeding
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group B (N=34) | IGB Group A (N=32)
surgical wound infection (Infections and infestations) | 8 (15) | 7 (9) — mild surgical wound infection ,mild respiratory failure ,eventration, intra abdominal abscess, urinary tract infection, bleeding, haematoma,pneumonia

LIMITATIONS AND CAVEATS:
we could not reach the number of scheduled patients in the study, due to the number of postrandomization excluded patients; the number of superobese is too short in order to get conclusion in this small group of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No